CLINICAL TRIAL: NCT00394381
Title: Autologous Cytokine-induced Killer Cell Adoptive Immunotherapy for Acute Myeloid Leukemia and Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIK#1/2006
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome, High Grade
Keywords: acute myeloid leukemia; myelodysplastic syndrome; autologous CIK cells; autologous peripheral blood stem cell transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CIK infusion (Experimental): Infusion of autologous CIK cells in study group. There is only one arm to this study
  Interventions: Procedure: Infusion of autologous CIK cells

INTERVENTIONS:
Procedure: Infusion of autologous CIK cells — Autologous CIK cells will be infused at timed intervals after autologous transplant for AML for group 1 patients, and with or without some cytoreduction treatment for group 2 patients

SUMMARY:
A phase I/II study to explore the feasibility and efficacy of autologous CIK cells in patients with acute myeloid leukemia (AML)/ high grade myelodysplastic syndrome (MDS)

1. Group 1: As adjuvant therapy in minimal residual disease state after autologous PBSCT.
2. Group 2: As an adoptive immunotherapy in untreated disease state when conventional therapy with curative intent is not applicable

DETAILED DESCRIPTION:
This is a Phase I /II study on the feasibility / efficacy of adoptive immunotherapy with autologous CIK cells for the following 2 groups of patients who have AML or high grade MDS :

1. Group 1 patients in minimal residual disease state post autologous peripheral blood stem cell transplant ( PBSCT ), and
2. Group 2 patients with untreated high grade MDS or AML, who are not fit for standard curative intent chemotherapy.

The CIK cells will be generated by leukapheresis from patients and cultured in GMP facilities. Four repeated infusions will be given for a target dose of 1x10e10 T cell per infusion.

Efficacy will be assessed by

1. Disease free survival compared to historical control in group 1 given CIK cells post autologous PBSCT as adjuvant immunotherapy (n=20 over 3 years), and
2. Effect on the peripheral or marrow leukemia cell load in group 2 patients given CIK cells as alternative therapy in place of chemotherapy (n=10).

ELIGIBILITY:
Inclusion Criteria:

1. For Group 1: AML or MDS post autologous peripheral blood or marrow stem cell transplant.
2. For Group 2: High grade MDS ( RAEB or RAEBIT ) or AML, whom the haematologist in charge has assessed and deemed unfit for chemotherapy with curative intent.Patients must have fairly stable white cell count requiring only low dose or no myelosuppressive medication
3. Patients must understand the trial nature of this treatment and accept the possible absence of benefit.

Exclusion Criteria:

1. uncontrolled infection
2. life expectancy less than 6 weeks.
3. Contraindication to undergo one session of leukapheresis for PBMNC harvesting

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
blood count changes | three months
T lymphocyte subsets | three months
T cell functions | 3 months
adverse reactions | 24 hour

SECONDARY OUTCOMES:
relapse rate | 5 year
survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Yeh-Ching Linn, MBBS, MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Linn YC, Lau LC, Hui KM. Generation of cytokine-induced killer cells from leukaemic samples with in vitro cytotoxicity against autologous and allogeneic leukaemic blasts. Br J Haematol. 2002 Jan;116(1):78-86. doi: 10.1046/j.1365-2141.2002.03247.x. PMID 11841399
- [Background] Leemhuis T, Wells S, Scheffold C, Edinger M, Negrin RS. A phase I trial of autologous cytokine-induced killer cells for the treatment of relapsed Hodgkin disease and non-Hodgkin lymphoma. Biol Blood Marrow Transplant. 2005 Mar;11(3):181-7. doi: 10.1016/j.bbmt.2004.11.019. PMID 15744236
- [Background] Schmidt-Wolf IG, Finke S, Trojaneck B, Denkena A, Lefterova P, Schwella N, Heuft HG, Prange G, Korte M, Takeya M, Dorbic T, Neubauer A, Wittig B, Huhn D. Phase I clinical study applying autologous immunological effector cells transfected with the interleukin-2 gene in patients with metastatic renal cancer, colorectal cancer and lymphoma. Br J Cancer. 1999 Nov;81(6):1009-16. doi: 10.1038/sj.bjc.6690800. PMID 10576658
- [Background] Jiang H, Liu KY, Tong CR, Jiang B, Lu DP. [The efficacy of chemotherapy in combination with auto-cytokine-induced killer cells in acute leukemia]. Zhonghua Nei Ke Za Zhi. 2005 Mar;44(3):198-201. Chinese. PMID 15840260